CLINICAL TRIAL: NCT06327373
Title: A Feasibility Study of Supplemental Oxygen to Improve Pulmonary Hypertension in People With Intradialytic Hypoxemia
Acronym: SOPHIE
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00114903
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Room air (Placebo Comparator): Participants will receive no supplemental oxygen.
  Interventions: Drug: Room air
- Supplemental oxygen (0.5 liters per minute) (Experimental): Participants will receive supplemental oxygen by oxygen concentrator delivered by nasal cannula at 0.5 liters per minute.
  Interventions: Drug: Oxygen
- Supplemental oxygen (3 liters per minute) (Experimental): Participants will receive supplemental oxygen by oxygen concentrator delivered by nasal cannula at 3 liters per minute.
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: Oxygen — Supplemental oxygen by oxygen concentrator
  Arms: Supplemental oxygen (0.5 liters per minute); Supplemental oxygen (3 liters per minute)
Drug: Room air — Room air without oxygen concentrator
  Arms: Room air

SUMMARY:
The purpose of this study is to assess the feasibility of supplemental oxygen delivery during hemodialysis in people with pulmonary hypertension and intradialytic hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years
* Receiving Monday-Wednesday-Friday or Tuesday-Thursday-Saturday hemodialysis
* Screened positive for pulmonary hypertension (defined by tricuspid regurgitant velocity [TRV] >2.5 m/s on echocardiography) and intradialytic hypoxemia (defined by spending ≥1/3 treatment with O2 saturation <90%) or hypoxemia for ≥10% of the treatment if associated with a desaturation event (≥4% decline in O2 saturation to <88% for ≥10 seconds) during enrollment in the PH-ESKD study (Pro00108710).

Exclusion Criteria:

* Daily supplemental oxygen use
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change daily hypoxemia burden | Weeks 1, 2, and 3
  Minutes with oxygen saturation <90% over a 24-hour period assessed by pulse oximetry

SECONDARY OUTCOMES:
Change in six minute walk distance | Weeks 1 and 3
  Scores are measured as meters walked during a six-minute assessment
Change in Montreal Cognitive Assessment (MoCA) | Weeks 1 and 3
  Scores are measured on a 30-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Edmonston, MD, MHS, Principal Investigator — Duke University
Locations (11):
- United States (11):
  - Davita Durham East, Durham, North Carolina
  - Davita Durham Downtown, Durham, North Carolina
  - Davita Research Triangle Park, Durham, North Carolina
  - Davita Durham Regional, Durham, North Carolina
  - Davita Durham West, Durham, North Carolina
  - Davita Bull City, Durham, North Carolina
  - Davita Durham Southpoint, Durham, North Carolina
  - Davita Hope Valley, Durham, North Carolina
  - Davita Vance County, Henderson, North Carolina
  - Davita Kerr Lake, Henderson, North Carolina
  - Davita Roxboro, Roxboro, North Carolina

IPD SHARING:
Plan to Share IPD: No